CLINICAL TRIAL: NCT00374738
Title: Effects of an Alternative Treatment for Military Sexual Trauma on PTSD Symptoms, Neurosteroids and Brain Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samueli Institute for Information Biology (Other)
Collaborators: Duke University (Other); Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NC181BO-1 (IRB #01012); DUHS Protocol No. 5023-05-10R2 (Other: Duke University Health System (DUHS))
Record Dates: First submitted 2006-09-07; First posted 2006-09-11 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Stress Disorders
Keywords: Guided Imagery for Trauma (GIFT); Posttraumatic Stress Disorder (PTSD); Military Sexual Trauma (MST); Military Sexual Trauma - related PTSD
MeSH Terms: conditions — Stress Disorders, Traumatic; Stress Disorders, Post-Traumatic; Military Sexual Trauma | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GIFT Intervention (Experimental): Guided Imagery for Trauma (GIFT)
  Interventions: Behavioral: Guided Imagery for Trauma (GIFT)
- Music Control (No Intervention): Relaxing Music Audio control; same music used in guided imagery, with no narrative voice.

INTERVENTIONS:
Behavioral: Guided Imagery for Trauma (GIFT) — Guided Imagery for Trauma (GIFT) - music and voice narration over a 12-week intervention. The control intervention included a relaxing music audio (the same music used in the guided imagery audio but without the narrative voiceover), PDA to log audio use, orientation and weekly phone consults, but did not have access to the patient advocate or to the guided imagery instructions provided on the GIFT audio.
  Arms: GIFT Intervention

SUMMARY:
Our specific aims are:

1. To examine the efficacy of GIFT in improving MST-related clinical outcomes in women veterans
2. To examine the effects of GIFT on fronto-limbic brain function and
3. To examine the effects of GIFT on levels of neuroactive steroid associated with PTSD.

DETAILED DESCRIPTION:
Guided imagery is a complementary and alternative treatment (CAM) modality. This directed meditation technique uses healing imagery to promote recovery in a variety of illnesses, including cancer, heart disease and, more recently, posttraumatic stress disorder (PTSD). PTSD is a severe and disabling anxiety disorder. It is among the most common mental disorders, affecting 10% of women in the United States during their lifetime. Sexual assault is the most common cause of PTSD. Similarly, military sexual trauma (MST) is disturbingly common among women in the armed forces. At least 20% of women veterans using VA services report a history of sexual assault. Unfortunately, high rates of MST-related PTSD are anticipated among women currently deployed to Iraq and Afghanistan.

To address this issue, we will evaluate a guided imagery intervention for women veterans who have MST-related PTSD. We will evaluate the efficacy of Guided Imagery for Trauma (GIFT) in decreasing PTSD symptoms. Using brain-imaging techniques, this research will examine the effects of GIFT on brain function in the areas associated with PTSD. We will also examine the effects of GIFT on neurosteroids, which are candidate modulators of PTSD symptoms, and may also represent novel targets for therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65
* Status as a woman veteran
* Receives care at the Durham VAMC
* History of MST
* DSM-IV diagnosis of PTSD, confirmed by CAPS interview
* Able to participate in a research interview in English
* Regular telephone access

Exclusion Criteria:

* Current diagnosis of organic or psychotic mental disorder
* Suicidality or parasuicidality
* Ongoing family violence
* Alcohol or drug dependence within previous 3 months
* Enrolled in cognitive-behavioral/exposure-based therapy during study period.
* Supportive therapy and psychiatric medications (if stabilized at least 3 months prior to enrollment) are acceptable.
* An uncontrolled medical condition

Exclusion Criteria for the fMRI only:

* Foreign metallic objects or implanted devices in the body incompatible with MRI
* Positive pregnancy test as determined by serum ß-HCG level
* Claustrophobia
* CNS neoplasms or neurological conditions such as Parkinson's Disease, Huntington's Chorea, demyelinating diseases, seizures, hydrocephalus, etc.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L. Strauss, PhD, Principal Investigator — Duke University Medical Center & Durham VA Medical Center; Christine Marx, MD, MA, Principal Investigator — Duke University Medical Center & Durham VA Medical Center
Locations (1):
- Women Veterans' Comprehensive Health Center (WVCHC) @ Durham Veterans Affairs Medical Center (DVAMC), Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Study terminated/inactive.